CLINICAL TRIAL: NCT05550779
Title: What Makes People Better at Retrieving Proper Names?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Colorado Springs (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Lori James, Professor, University of Colorado, Colorado Springs
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2023-023; R15AG063111-01 (NIH)
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy Aging
Keywords: cognitive aging; name retrieval

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two mental exercises before performing a proper name production task and completing other measures.
Who Masked: Participant
Masking Description: Participants do not know which condition they are in, nor that there is another condition. They only know what mental exercise they will do in their assigned condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Exercise A (Experimental): Participants follow instructions on a 10-minute audio clip
  Interventions: Behavioral: Mental Exercise
- Mental Exercise B (Active Comparator): Participants follow instructions on a 10-minute audio clip
  Interventions: Behavioral: Mental Exercise

INTERVENTIONS:
Behavioral: Mental Exercise — Participant perform a 10-minute mental exercise

SUMMARY:
This study is being conducted to learn more about how various personal and situational characteristics are related to the ability to produce names of pictured people. Participants will perform a brief mental exercise, then see 83 celebrity photographs to produce the names of. Participants will also complete other surveys and measures. Collected data will give researchers a better understanding of how different variables relate to proper name production.

DETAILED DESCRIPTION:
This study is being conducted to learn more about how various personal and situational characteristics are related to the ability to produce names of pictured people. Adult participants ages 18-35 and 60-80 will participant in videoconference calls during which they will perform a brief mental exercise, then see 83 celebrity photographs with instructions to name each pictured person. The naming task will be video recorded for later scoring. Participants will also complete other surveys and measures, including some about demographics and other personal characteristics. Participation will take approximately 60-75 minutes. Collected will be de-identified and the aggregate data will give researchers a better understanding about how individual's personality and cognitive traits and the mental exercise performed before the study relate to people's proper name production.

ELIGIBILITY:
Inclusion Criteria:

* fluent speaker of English
* ages 18-35 or 60-80
* lived in the United States for at least 5 years

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori James, PhD, Principal Investigator — University of Colorado, Colorado Springs
Locations (1):
- UCCS, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
De-identified participant data may be posted on a website for open access to other researchers, if the publication outlet requires it. But I do not currently plan to share the data

RESULTS

PARTICIPANT FLOW:
Groups:
- Mental Exercise: Intervention: Participants follow instructions on a 10-minute audio clip with mindful breathing
  Mental Exercise: Participant perform a 10-minute mental exercise
- Mental Exercise: Control: Participants follow instructions on a 10-minute audio clip about a story
  Mental Exercise: Participant perform a 10-minute mental exercise
Period: Overall Study
Arm/Group | Mental Exercise: Intervention | Mental Exercise: Control
Started | 54 | 55
Completed | 54 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mental Exercise: Control: Participants follow instructions on a 10-minute audio clip of a story
  Mental Exercise: Participant perform a 10-minute mental exercise
- Total: Total of all reporting groups
Arm/Group | Mental Exercise: Intervention | Mental Exercise: Control | Total
Number analyzed (Participants) | 54 | 55 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 28 | 56
  >=65 years | 26 | 27 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 46 | 87
  Male | 13 | 9 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 52 | 52 | 104
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 41 | 43 | 84
  More than one race | 4 | 4 | 8
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent of Familiar Faces With TOT Responses
Description: Percent of trials with name retrieval failures were measured on a task created for this purpose. Specifically, participants tried to provide names that fit photographs, indicating when a name got stuck on the "tip of their tongue" by saying "TOT."
Time Frame: During the 60-75 minute experimental session
Population: Some participants completed the experiment but their data were not included due to having distractions present during testing (e.g., another individual interrupting the participant), experiencing a terrible internet connection during testing, being uncomfortable with turning on their video during testing, and not meeting the age inclusion criteria after initially claiming that they did.
Measure: Mean (Standard Deviation); unit: Percent of familiar faces with TOTs
Groups:
- Mental Exercise: Intervention: Participants follow instructions on a 10-minute audio clip of mindful breathig
  Mental Exercise: Participant perform a 10-minute mental exercise
Arm/Group | Mental Exercise: Intervention | Mental Exercise: Control
Number analyzed (Participants) | 51 | 51
Percent of familiar faces with TOTs
  Young Adults: number analyzed (Participants) | 26 | 25
  Young Adults | 16 (14) | 15 (9)
  Older Adults: number analyzed (Participants) | 25 | 26
  Older Adults | 18 (14) | 15 (12)

2. Primary Outcome: Percent of Known Names With TOT Responses
Description: Percent of trials with name retrieval failures were measured on a task created for this purpose. Specifically, participants tried to provide names that fit photographs, indicating when a name got stuck on the "tip of their tongue" by saying "TOT." These percentages are out of correct and TOT responses only.
Time Frame: During the 60-75 minute experimental session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of known names with TOTs
Arm/Group | Mental Exercise: Intervention | Mental Exercise: Control
Number analyzed (Participants) | 51 | 51
Percent of known names with TOTs
  Young Adults: number analyzed (Participants) | 26 | 25
  Young Adults | 15 (9) | 16 (14)
  Older Adults: number analyzed (Participants) | 25 | 26
  Older Adults | 15 (12) | 18 (14)

3. Primary Outcome: Percent of Unknown Names With TOT Responses
Description: Percent of trials with name retrieval failures were measured on a task created for this purpose. Specifically, participants tried to provide names that fit photographs, indicating when a name got stuck on the "tip of their tongue" by saying "TOT." These percentages are out of all responses that are not correct or TOTs only.
Time Frame: During the 60-75 minute experimental session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of unknown names with TOTs
Arm/Group | Mental Exercise: Intervention | Mental Exercise: Control
Number analyzed (Participants) | 51 | 51
Percent of unknown names with TOTs
  Young Adults: number analyzed (Participants) | 26 | 25
  Young Adults | 41 (22) | 37 (25)
  Older Adults: number analyzed (Participants) | 25 | 26
  Older Adults | 39 (25) | 34 (20)

ADVERSE EVENTS:
Time Frame: 1.25 hour experimental session
Description: This minimal-risk, brief behavioral intervention poses almost no risk, and certainly no serious risk of adverse events.
Arm/Group | Mental Exercise: Intervention | Mental Exercise: Control
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/55
Other Adverse Events (participants affected / at risk) | 0/54 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-09-05): https://cdn.clinicaltrials.gov/large-docs/79/NCT05550779/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-05): https://cdn.clinicaltrials.gov/large-docs/79/NCT05550779/SAP_001.pdf
  • Informed Consent Form (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT05550779/ICF_002.pdf